CLINICAL TRIAL: NCT03315065
Title: Feasibility Study to Determine Utility of 19F MRI for Regional Pulmonary Function Assessment in Patients Receiving Thoracic Radiotherapy for Lung Cancer
Brief Title: 19F Thoracic Radiotherapy for Lung Cancer
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Hal C Charles (Other)
Responsible Party: Sponsor-Investigator, Hal C Charles, Associate Professor Radiology, Duke University
Organization: Duke University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00084472
Record Dates: First submitted 2017-10-11; First posted 2017-10-19 (Actual); Last update posted 2019-07-16 (Actual); Status verified 2019-07

CONDITIONS: Lung Cancer
Keywords: thoracic Radiation therapy; Lung Function
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Patients diagnosed with Lung cancer (Other): patients diagnosed with Lung cancer and Thoracic radiotherapy
  Interventions: Drug: Perfluorinated Gas/Oxygen Mixture

INTERVENTIONS:
Drug: Perfluorinated Gas/Oxygen Mixture — 19-Fluorine (19F) MRI of the lungs with 21%/79% Oxygen/Perfluorinated Gas, ≤ 25 liters, gas and Mixture of 30% perfluoropropane and 70% oxygen to measure perfusion single visit, < 1 hour
  Other Names: Perfluorinated Propane Imaging

SUMMARY:
The goal of this study is to determine the feasibility and efficiency of incorporating 19F MR functional lung imaging into the routine assessment of lung cancer patients prior to thoracic radiotherapy.

DETAILED DESCRIPTION:
Primary Objective:

Determine feasibility by evaluating if:

PO1: Patients diagnosed with lung cancer are able to successfully complete pre- and post-radiotherapy 19F MR imaging scans as scheduled.

Secondary Objective:

Determine efficiency by evaluating if:

SO1: Determine efficiency by evaluating if 19F MRI data can be successfully analyzed and incorporated into the radiation planning system.

SO2: Determine efficiency by evaluating if the incorporated 19F MRI functional data can be successfully used to generate radiotherapy plan in a timely manner.

SO3: Determine if pre- and post radiotherapy 19F MRI scans can be readily compared to observe changes in pulmonary function.

Hypotheses Investigators hypothesize that functional 19F MR imaging assessment is feasible in the lung cancer patient population and that the acquired images can be efficiently analyzed and integrated into radiotherapy planning.

ELIGIBILITY:
Inclusion Criteria:

* Subject has histologic or cytologic confirmation of lung cancer (NSCLC or Small cell) and has been recommended thoracic radiotherapy as part of standard of care management.
* Ability to undergo MR imaging, tolerate breath hold procedures and follow direction during the imaging process
* Karnofsky performance status ≥60, with expected survival of ≥6 months
* At least 18 years of age
* Patient is not pregnant
* Patient can be reliably reached for post-MRI follow up AE check.
* Patient able to sign a study specific informed consent form.

Exclusion Criteria:

* Any condition including, metallic implants or cardiac pacemakers that makes the candidate ineligible for MR imaging. (MRI research screening form will be completed prior to each MRI scan).
* Malignant pleural effusion or pericardial effusion

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-02-16 (Actual); Primary Completion 2019-06-25 (Actual); Study Completion 2019-06-25 (Actual)

PRIMARY OUTCOMES:
Number of study patients consented (maximum 8)in order to result in 5 patients successfully completing both 19F functional MR imaging data sets | 4 months
Proportion of study patients that successfully return for a re-assessment 19F MRI scan after completing radiotherapy. | 6 weeks after completing RT

CONTACTS AND LOCATIONS:
Overall Officials: Kolby Sidhu, MD, Principal Investigator — Duke University Medical Center, Department of Radiation Oncology
Locations (1):
- Duke University Medical Center - Cancer Center, Durham, North Carolina, United States